CLINICAL TRIAL: NCT03228459
Title: Randomized Intervention Study to Assess the Prevalence of Subclinical Vascular Disease and Hidden Kidney Disease and Its Impact on Morbidity and Mortality: The ILERVAS Project
Brief Title: The ILERVAS Project: Assessing the Prevalence of Subclinical Vascular Disease and Hidden Kidney Disease
Acronym: ILERVAS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut de Recerca Biomèdica de Lleida (Other)
Collaborators: Diputació de Lleida (Unknown); Jaume Arnó Renal Foundation (Other); Unit of Detection and Treatment of Atherothrombotic diseases (UDETMA) (Unknown); Lleida Primary health care (Unknown)
Responsible Party: Principal Investigator, Elvira Fernández Giráldez, Study Chair, Institut de Recerca Biomèdica de Lleida
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: The ILERVAS project
Record Dates: First submitted 2017-07-17; First posted 2017-07-25 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Atherosclerosis; Chronic Kidney Diseases; Metabolic Syndrome; PreDiabetes; Subclinical Disease and/or Syndrome
Keywords: Kidney Diseases; Subclinical Disease and/or Syndrome; Atherosclerosis; Biomarkers; Prevention; Lung capacity; Early diagnosis; Advanced glycation-end products; Atrial fibrillation; Diabetes; Arterial ultrasound
MeSH Terms: conditions — Atherosclerosis; Renal Insufficiency, Chronic; Metabolic Syndrome; Prediabetic State; Kidney Diseases; Disease; Atrial Fibrillation; Diabetes Mellitus | interventions — Urinalysis; Ultrasonography, Carotid Arteries; Ankle Brachial Index; Spirometry; Pulse Wave Analysis

STUDY DESIGN:
Intervention Model Description: A randomized interventional study with 2 arms that will include 16,660 individuals with at least one cardiovascular risk factor from the province of Lleida, Spain. Patients will be recruited from January 2015 to December 2018. Patients will be followed for 10 years.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mobile Unit Follow-up Group (Experimental): In the Mobile Unit (MU), clinical, sociodemographic and anthropometric data will be recorded. Patients will be evaluated with artery ultrasound (carotid, femoral, transcranial and abdominal aorta), ankle-brachial index, pulse wave velocity, spirometry, determination of advanced glycation-end products, atrial fibrillation screening, dried blood spot test and urine analysis. Moreover, DNA, RNA, Saliva, blood and urine samples will be collected and stored in the biobank to identify new biomarkers using omic studies. Additionally, climate, air pollutant and airborne pollen data form the entire province of Lleida will be registered. Finally, a report with the exploration results and recommendations based on the current guidelines will be uploaded to the e-CAP history for the Primary care evaluation.
  Interventions: Diagnostic Test: Dried blood spot test; Diagnostic Test: Urine test; Diagnostic Test: Artery ultrasound; Diagnostic Test: Ankle-brachial index; Diagnostic Test: Spirometry; Diagnostic Test: Determination of advanced glycation-end products; Diagnostic Test: Atrial fibrillation screening; Other: Biological sample collection; Other: Result and recommendation report; Diagnostic Test: Pulse wave velocity
- Electronic Medical History Follow-up Group (No Intervention): Participants will be followed through their electronic medical records. Sociodemographic (age, sex, race, marital status, education and labour status), clinical and anthropometric data and will be electronically collected.

INTERVENTIONS:
Diagnostic Test: Dried blood spot test — Dried capillary blood testing creatinine, uric acid and total cholesterol (reflotron® Plus system, Roche). Determination of the complete lipid profile in cases in which total cholesterol is greater than 200 mg/dl: HDL cholesterol (mg/dl), LDL cholesterol (mg/dl) and triglycerides (mg/dl) (Cobas B 101® system, Roche). Calculation of non-HDL cholesterol levels. Glycated haemoglobin will be analysed with the Cobas B 101 system,Roche. The CKD-EPI glomerular filtration rate will be determined.
  Arms: Mobile Unit Follow-up Group
Diagnostic Test: Urine test — A urine sample from spontaneous micturition will be collected and analyzed using Clinitek Microalbumin 2 Reagent Strips and a Siemens Clinitek Status® analyzer. It will be determined albuminuria (mg/l) and albumin/creatinine ratio (mg/g).
  Arms: Mobile Unit Follow-up Group
Diagnostic Test: Artery ultrasound — Carotid and femoral artery ultrasound for atheroma plaque diagnosis. Abdominal aorta ultrasound for early diagnosis of aortic aneurism. Transcranial ultrasound for cerebral arterial blood flow alterations.
  Arms: Mobile Unit Follow-up Group
Diagnostic Test: Ankle-brachial index — Systolic blood pressure measurement in the brachial artery, posterior tibial artery and dorsalis pedis artery in both limbs. The ratios between tibial and pedal systolic blood pressure in each leg and the higher brachial blood pressure will be calculated.
  Arms: Mobile Unit Follow-up Group
Diagnostic Test: Spirometry — Spirometry will be used to assess lung capacity. It will be performed by the same nurse who will measure forced vital capacity (FVC); forced expiratory volume in one second (FEV1); the ratio between FEV1 and FVC and the lower limit of normality, as a percentage.
  Arms: Mobile Unit Follow-up Group
Diagnostic Test: Determination of advanced glycation-end products — These will be measured using skin autofluorescence (SAF) in the forearm with the AGE Reader® system (Diagnostics, the Netherlands). SAF is measured using spectrophotometry which is calculated as the relationship of the intensity of reflected light compared to refracted light.
  Arms: Mobile Unit Follow-up Group
Diagnostic Test: Atrial fibrillation screening — The presence of atrial fibrillation is assessed with a device (SRA, EVINA Health Solutions) during one hour in the mobile unit.
  Arms: Mobile Unit Follow-up Group
Other: Biological sample collection — Blood samples from a peripheral vein of the hand or forearm to obtain serum, plasma, DNA and RNA will be collected. Moreover, a saliva sample will be collected.These samples will be prepared in aliquots following a standardized protocol, and sent frozen (dry ice) to a centralized biobank (IRBLleida Biobank, Spain) for processing and storage for subsequent studies of CV, inflammatory and mineral-metabolism biomarkers and genetic polymorphisms. Urine samples will be frozen and stored in a biobank for subsequent study of biomarkers.
  Arms: Mobile Unit Follow-up Group
Other: Result and recommendation report — A report with exploration results and recommendations based on the current guidelines will be uploaded to the e-CAP history for the Primary care evaluation.
  Arms: Mobile Unit Follow-up Group
Diagnostic Test: Pulse wave velocity — Pulse wave velocity (PWV) will be used as an indicator of arterial stiffness. It will be measured non-invasively with the carotid to femoral PWV (cfPWV) according to standard protocols.
  Arms: Mobile Unit Follow-up Group

SUMMARY:
BACKGROUND AND OBJECTIVES:

Cardiovascular disease is the leading cause of death despite huge primary and secondary prevention policies with a strong economic burden. The primary objectives of the ILERVAS project are: (i) to identify unknown factors involved in the presence of atherosclerosis, metabolic syndrome, pre-diabetes and hidden kidney disease in a low/moderate cardiovascular risk population; (ii) to identify unknown factors involved in the progression of atherosclerosis, metabolic syndrome, pre-diabetes and hidden kidney disease in a low/moderate cardiovascular risk population; (iii) to Assess of the impact of arterial ultrasound on cardiovascular events and mortality in a low/moderate cardiovascular risk population.

METHODS:

Randomized intervention study. From 2015 to 2018, 16,660 participants (8,330 in the intervention group (Mobile Unit Follow-up Group) and 8,330 in the no intervention group (Electronic Medical History Follow-up Group )) aged between 45 and 70 years without a previous history of cardiovascular disease and with at least one cardiovascular risk factor will be randomly selected across the province of Lleida, Spain.

DETAILED DESCRIPTION:
STUDY DESIGN AND POPULATION:

Randomized interventional study. From 2015 to 2018, 16,660 participants (8,330 in the intervention group (Mobile Unit Follow-up Group) and 8,330 in the no intervention group (Electronic Medical History Follow-up Group)) aged between 45 and 70 years without a previous history of cardiovascular disease and with at least one cardiovascular risk factor will be randomly selected across the province of Lleida, Spain. The Ethics Committee of the University Hospital Arnau de Vilanova in Lleida (Spain) approved the protocol. All patients signed informed consent. The study was conducted according to the principles of the Declaration of Helsinki.

SOURCE OF INFORMATION AND INSTRUMENTS FOR DATA COLLECTION:

In the Mobile Unit (MU), clinical, sociodemographic and anthropometric data will be recorded. Patients will be evaluated with artery ultrasound (carotid, femoral, transcranial and abdominal aorta), ankle-brachial index, pulse wave velocity, spirometry, determination of advanced glycation-end products, atrial fibrillation screening, dried blood spot test and urine analysis. Moreover, DNA, RNA, Saliva, blood and urine samples will be collected and stored in the biobank to identify new biomarkers using omic studies. Additionally, climate, air pollutant and airborne pollen data form the entire province of Lleida will be registered. In addition, variables such as physical exercise, diet and daytime will be collected.

In the no intervention group (Electronic Medical History Follow-up Group), participants will be followed through their electronic medical records. Sociodemographic (age, sex, race, marital status, education and labour status), clinical and anthropometric data and will be electronically collected.

PARTICIPANT SELECTION:

From a total of 410,246 people with an open history in the e-CAP (in October 24, 2014), the study population that meets the inclusion criteria will be identified. Of these, a total of 16,660 people (8,330 in the intervention group and 8,330 in the no intervention group) will be selected through simple randomization without replacement, within clusters defined by basic healthcare area, primary care (PC) centre or doctor's office, in accordance with the total number of people who may be visited in the MU during one year period. The participants of the selected intervention group will be informed of the study objectives and the diagnostic tests.

FOLLOW-UP PERIOD:

A minimum 10-year follow-up period has been established to observe the onset of CV events. In the Mobile Unit Follow-up group, a second visit will be performed after four year of recruitment.

CARDIOVASCULAR EVENTS AND CKD PROGRESSION:

The onset of a CV event will be recorded according to the 10th version of the International Statistical Classification of Diseases (ICD-10), which includes: angina pectoris, myocardial infarction, transient ischemic attack, cerebrovascular accident, heart failure, arrhythmia, peripheral artery disease, aortic aneurysm, revascularization and angioplasty of any artery region. Likewise, the patient's cause of death, whether of CV origin (myocardial infarction, arrhythmia, heart failure, cerebrovascular accident, aortic aneurysm, mesenteric infarction or sudden death) or of non-CV origin (infections, cancers, accident or kidney disease) will be recorded. The information sources used to identify CV events will be: review of medical records (through the e-CAP) and consultation of the Catalonia mortality registry. CKD progression is defined as a doubling of creatinine or entry into renal replacement therapy, and will also be collected through the e-CAP.

CLINICAL AND BIOCHEMICAL DATA:

The following variables will be recorded: weight, height, waist circumference and neck circumference, body mass index in kg/m2, hours of fasting, systolic blood pressure, diastolic blood pressure and pulse pressure (mmHg). Blood pressure will be measured 3 times (Omron 6®) at 2-min intervals and the mean of the last 2 will be collected. Dried capillary blood testing (fingertip puncture) will be used to determine creatinine, uric acid and total cholesterol, using the reflotron® Plus system (Roche). In cases in which total cholesterol is greater than 200 mg/dl, the complete lipid profile (HDL cholesterol, LDL cholesterol and triglycerides) will be determined using Cobas B 101® system, Roche. Non-HDL cholesterol levels, glycated hemoglobin (Cobas B 101 system, Roche), the CKD-EPI glomerular filtration rate will be determined as well. Albuminuria and albumin/creatinine ratio will be determined in urine sample from spontaneous micturition collected in the MU using Clinitek Microalbumin 2 Reagent Strips and a Siemens Clinitek Status® analyzer.

ARTERY ULTRASOUND:

The examination and reading will be performed by 2 nurses specialized in vascular imaging diagnostics, following a standardized protocol with the patient in supine decubitus. The VIVID I version BT12 ultrasound system (GE Healthcare) will be used. The system has a 12L-RS/4-13 MHz linear probe (carotid and femoral arteries), a 4C-RS/1.5-6 MHz convex probe (abdominal aorta) and a 3SRS/ 1.5-2.5 MHz sector probe (transcranial). It also has a module for measuring intima-media thickness and pulsed Doppler ultrasound to assess hemodynamic abnormalities in the case that atheromatous plaques are present, and also to analyze the intracranial circulation. The DICOM network connectivity system will be used to record the results and ultrasound images online in the e-CAP.

Carotid arteries: a total of 8 vascular regions will be analyzed (common carotid, bifurcation or bulb, internal carotid and external carotid), with the patient in supine decubitus and the head turned 45º towards the opposite side in the examination.

Femoral arteries: with the patient in supine decubitus, the presence of plaque will be examined in the common femoral artery (1 cm proximal to the bifurcation) and the superficial femoral artery on both sides. The plaque definition follows the same previous criteria.

Abdominal aorta: in men age 60 and older. With the patient in supine decubitus, the abdominal aorta will be examined in the midline of the abdomen from the base of the sternum until the bifurcation the iliac arteries. In an axial section, at the points where a greater diameter is observed, 2 images of the aorta will be captured, and 2 measurements will be made (anterior-posterior and lateral-lateral). An aortic aneurysm will be considered to be present when the diameter is greater than 3 cm.

Transcranial ultrasound: the arteries of the Willis circle and their branches will be insonated through the transtemporal and transforaminal acoustic windows. The Doppler spectrum of each intracranial artery will be determined using the colour-coded signal. Flow direction, peak systolic velocity, mean flow velocity and diastolic flow velocity will be established. The intracranial carotid artery, the medial cerebral artery in the M1 and M2 segments, the anterior cerebral artery (segment A1) and the posterior cerebral artery in segments P1 and P2 will be studied through the transtemporal acoustic window. The V4 segment of the vertebral arteries and the basilar artery will be studied through the transforaminal acoustic window. In each patient, the number, location and severity of stenosis will be recorded. Baumgartner's criteria will be used to establish the severity of the stenosis based on peak systolic wave velocity (moderate to serious stenosis, if it is ≥155/ 220 cm/s for the medial cerebral artery, ≤120/≥155 cm/s for the anterior cerebral artery, ≥100/≥145 cm/s for the posterior cerebral artery and the basilar artery, and ≥90/≥120 cm/s for the vertebral artery).

ANKLE-BRACHIAL INDEX:

A continuous Doppler (Hadecco ES100X MiniDop®), sphygmomanometer and blood pressure cuffs (Riester minimus III®) will be used. Systolic blood pressure will be measured in the brachial artery, posterior tibial artery and dorsalis pedis artery in both limbs. The ratios between tibial and pedal systolic blood pressure in each leg and the higher brachial blood pressure will be calculated. The final value for each limb will be the lower value of those obtained between tibial and pedal blood pressure. An ankle-brachial index value <0.9 will be considered to be suggestive of stenosis; a value <0.7 will be considered to be stenosis and a value ≥1.4 will be considered to be suggestive of arterial rigidity.

SPIROMETRY:

Spirometry will be used to assess lung capacity. It will be performed by the same nurse who will measure forced vital capacity (FVC); forced expiratory volume in one second (FEV1); the ratio between FEV1 and FVC and the lower limit of normality, as a percentage.

DETERMINATION OF ADVANCED GLYCATION-END PRODUCTS:

They will be measured using skin autofluorescence (SAF) in the forearm with the AGE Reader system® (Diagnostics, the Netherlands). SAF is measured using spectrophotometry which is calculated as the relationship of the intensity of reflected light compared to refracted light. The result obtained will be divided into 4 CV risk groups, taking into account age and sex.

ATRIAL FIBRILLATION SCREENING:

The presence of atrial fibrillation will be assessed with the SRA device® (EVINA Health Solutions) for one hour in the MU.

PULSE WAVE VELOCITY:

Pulse wave velocity (PWV) will be used as an indicator of arterial stiffness. It will be measured non-invasively with the carotid to femoral PWV (cfPWV) according to standard protocols.

BIOLOGICAL SAMPLE COLLECTION:

Blood samples from a peripheral vein of the hand or forearm to obtain serum, plasma, DNA and RNA will be collected. Moreover, a saliva sample will be collected.These samples will be prepared in aliquots following a standardized protocol, and sent frozen (dry ice) to a centralized biobank (IRBLleida Biobank, Spain) for processing and storage for subsequent studies of CV, inflammatory and mineral-metabolism biomarkers and genetic polymorphisms. Urine samples will be frozen and stored in a biobank for subsequent study of biomarkers.

STATISTICAL ANALYSIS:

Descriptive analysis will include absolute and relative frequencies for the qualitative variables, means and standard deviations for the continuous variables that follow a normal distribution, and median and interquartile range in the cases that do not follow a normal distribution. Their distribution will be analyzed with the chi-squared test, in the case of qualitative variables, and Student's t test or ANOVA for quantitative variables with a normal distribution, or, failing this, non-parametric Mann-Whitney U or Kruskal-Wallis tests will be used for those without a normal distribution. The correlation between quantitative variables will be analyzed using Pearson's or Spearman's test, depending on the distribution. The existence of collinearity between 2 variables will be analyzed to enter the variable that better predicts the result variable in the multivariate model. Multivariate analysis will be performed using logistic regression if the dependent variable is qualitative or linear regression if it is quantitative. Beta regression coefficients, odds ratios (ORs) and their respective 95% confidence intervals will be estimated as measures of association. In the longitudinal study, the incidence of CV morbidity and mortality and mortality due to any cause will be analyzed, based on the diagnostic tests used in the MU and the biomarkers studied using Cox regression. Statistical significance will be set at a p value < 0.05.

ELIGIBILITY:
Inclusion Criteria:

* women (50-70 years) and men ( 45-65 years) with at least one cardiovascular risk factor (hypertension, dyslipidemia, obesity (BMI >30 Kg/m2), current smoking habit or former smoker (<10 years), first-degree family history of early cardiovascular disease).

Exclusion Criteria:

* Prior medical history of cardiovascular disease.
* Diabetes.
* Glomerular filtration rate (CKD-EPI < 60 ml/min/1.73m2).
* Active neoplasm or acute disease.
* A life expectancy < 18 months.
* Pregnancy.

Ages: 45 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16660 (Actual)
Dates: Start 2015-01-15 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Identification of sociodemographic, lifestyle, clinical, anthropometric, laboratory, climate and air pollutants factors involved in atherosclerosis, in a low/moderate cardiovascular risk population. | 4 years
  The presence of atherosclerosis will be identified as an intima-media thickness higher than 1.5 mm.
Identification of sociodemographic, lifestyle, clinical, anthropometric, laboratory, climate and air pollutants factors involved in pre-diabetes, in a low/moderate cardiovascular risk population. | 4 years
  The percentage of glycated hemoglobin (Hb A1c) will be determined with a Cobas b 101® machine (Roche). Values lower than 5.7% are normal, > 5.7-6.5% indicate pre-diabetes; and ≥ 6.5% indicate diabetes.
Identification of sociodemograpic, lifestyle, clinical, anthropometric, laboratory, climate and air pollutants factors involved in chronic kidney disease, in a low/moderate cardiovascular risk population. | 4 years
  The prevalence of hidden chronic kidney disease will be assessed with a urine spot test that determines the albumin/creatinine ratio (ACR). Values lower than 30 mg/g are normal; 30-300 mg/g indicate microalbuminuria; and values higher than 300 indicate macroalbuminuria.
Assessment of the impact of arterial ultrasound on cardiovascular events and mortality in a low/moderate cardiovascular risk population. | 10 years
  The onset of a cardiovascular event will be recorded according to the tenth version of the International Statistical Classification of Diseases (ICD-10). Cardiovascular events and mortality in the intervention group will be compared to the control group during a during a 10-year follow-up period.

SECONDARY OUTCOMES:
Prevalence of atherosclerosis in a low/moderate cardiovascular risk population | 4 years
  The presence of atherosclerosis will be identified as an intima-media thickness higher than 1.5 mm.
Prevalence of hidden chronic kidney disease in a low/moderate cardiovascular risk population. | 4 years
  The prevalence of hidden chronic kidney disease will be assessed with a urine spot test that determines the albumin/creatinine ratio (ACR). Values lower than 30 mg/g are normal; 30-300 mg/g indicate microalbuminuria; and values higher than 300 indicate macroalbuminuria.
Prevalence of pre-diabetes and undiagnosed diabetes in a low/moderate cardiovascular risk population. | 4 years
  The percentage of glycated hemoglobin (Hb A1c) will be determined with a Cobas b 101® machine (Roche). Values lower than 5.7% are normal; 5.7-6.5% indicate pre-diabetes; and ≥ 6.5% indicate diabetes.
Correlation of skin autofluorescence with atherosclerosis in a low/moderate cardiovascular risk population. | 4 years
  Skin autofluorescence will be analyzed with the AGE reader™ device (DiagnOptics Technologies, Groningen, The Netherlands). Values range from 1-24 units.
Correlation of adherence to the Mediterranean diet with atherosclerosis in a low/moderate cardiovascular risk population. | 4 years
  Adherence to the Mediterranean diet will be evaluated with the Mediterranean Diet Adherence screener (MEDAS). Values are from 0 to 14 and categorize subjects according to their level of adherence: high (score >11 points), moderate (7-10 points), and low (<6 points).
Correlation of physical exercise with atherosclerosis in a low/moderate cardiovascular risk population. | 4 years
  Physical exercise will be evaluated with the International Physical Activity Questionnaire (IPAQ). Values are from vigorous, moderate, and low physical activity. Low activity corresponds to no activity or some activity but not enough to meet moderate category. Moderate corresponds to 3 or more days of walking for at least 30 minutes. Vigorous activity corresponds to 5 or more days of walking for at least 60 minutes.
Prevalence of atrial fibrillation in a low/moderate cardiovascular risk population. | 4 years
  The presence of atrial fibrillation is assessed with stroke risk analysis device (SRA, EVINA Health Solutions).
Correlation of spirometry alterations with atherosclerosis in a low/moderate cardiovascular risk population | 4 years
  Forced vital capacity (FVC) will be measured as liters (l).
Correlation of advanced glycation end-products (AGEs) and cardiovascular events in a low/moderate cardiovascular risk population. | 10 years
  AGES will be analyzed with the AGE reader™ device (DiagnOptics Technologies, Groningen, The Netherlands). Values range from 1-24 units.
Correlation of adherence to the Mediterranean diet and cardiovascular events in a low/moderate cardiovascular risk population. | 10 years
  Adherence to the Mediterranean diet will be evaluated with the Mediterranean Diet Adherence screener (MEDAS). Values are from 0 to 14 and categorize subjects according to their level of adherence: high (score >11 points), moderate (7-10 points), and low (<6 points).
Correlation of physical exercise and cardiovascular events in a low/moderate cardiovascular risk population. | 10 years
  Physical exercise will be evaluated with the International Physical Activity Questionnaire (IPAQ). Values are from vigorous, moderate, and low physical activity.
Association of spirometry alterations and cardiovascular events in a low/moderate cardiovascular risk population | 10 years
  Forced vital capacity (FVC) will be measured as liters (l).

CONTACTS AND LOCATIONS:
Overall Officials: Elvira Fernández Giráldez, MD, PhD, Study Chair — Fundació Renal Jaume Arnò; Marcelino Bermúdez López, MD, PhD, Study Director — Institut de Recerca Biomèdica de Lleida
Locations (3):
- Spain (3):
  - Fundació Renal Jaume Arnò, Lleida
  - Primary Care centre, Lleida
  - Institut de recerca Biomèdica de Lleida, Lleida

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Betriu A, Farras C, Abajo M, Martinez-Alonso M, Arroyo D, Barbe F, Buti M, Lecube A, Portero M, Purroy F, Torres G, Valdivielso JM, Fernandez E. Randomised intervention study to assess the prevalence of subclinical vascular disease and hidden kidney disease and its impact on morbidity and mortality: The ILERVAS project. Nefrologia. 2016 Jul-Aug;36(4):389-96. doi: 10.1016/j.nefro.2016.02.008. Epub 2016 Apr 1. English, Spanish. PMID 27044887
- [Result] Sanchez E, Lecube A, Betriu A, Hernandez C, Lopez-Cano C, Gutierrez-Carrasquilla L, Kerkeni M, Yeramian A, Purroy F, Pamplona R, Farras C, Fernandez E, Barbe F, Simo R; ILERVAS project; Hernandez M, Rius F, Polanco D, de la Torre MS, Torres G, Godoy P, Portero-Otin M, Jove M, Colas-Compas L, Benabdelhak I, Miquel E, Ortega M, Valdivielso JM, Bermudez M, Martinez-Alonso M. Subcutaneous advanced glycation end-products and lung function according to glucose abnormalities: The ILERVAS Project. Diabetes Metab. 2019 Dec;45(6):595-598. doi: 10.1016/j.diabet.2018.04.002. Epub 2018 Apr 13. No abstract available. PMID 29706471
- [Result] Montserrat-Capdevila J, Seminario MA, Godoy P, Marsal JR, Ortega M, Pujol J, Castan MT, Alseda M, Betriu A, Lecube A, Portero M, Purroy F, Valdivielso JM, Barbe F. Prevalence of chronic obstructive pulmonary disease (COPD) not diagnosed in a population with cardiovascular risk factors. Med Clin (Barc). 2018 Nov 21;151(10):383-389. doi: 10.1016/j.medcli.2017.12.018. Epub 2018 Mar 7. English, Spanish. PMID 29525115
- [Result] Gutierrez-Carrasquilla L, Sanchez E, Hernandez M, Polanco D, Salas-Salvado J, Betriu A, Gaeta AM, Carmona P, Purroy F, Pamplona R, Farras C, Lopez-Cano C, Fernandez E, Lecube A. Effects of Mediterranean Diet and Physical Activity on Pulmonary Function: A Cross-Sectional Analysis in the ILERVAS Project. Nutrients. 2019 Feb 3;11(2):329. doi: 10.3390/nu11020329. PMID 30717453
- [Result] Sanchez E, Betriu A, Yeramian A, Fernandez E, Purroy F, Sanchez-de-la-Torre M, Pamplona R, Miquel E, Kerkeni M, Hernandez C, Simo R, Lecube A; ILERVAS project; ILERVAS Project:; Hernandez M, Rius F, Polanco D, Barbe F, Torres G, Suarez G, Portero-Otin M, Jove M, Colas-Campas L, Benabdelhak I, Farras C, Ortega M, Manuel Valdivielso J, Bermudez-Lopez M, Martinez-Alonso M. Skin Autofluorescence Measurement in Subclinical Atheromatous Disease: Results from the ILERVAS Project. J Atheroscler Thromb. 2019 Oct 1;26(10):879-889. doi: 10.5551/jat.47498. Epub 2019 Mar 6. PMID 30842389
- [Result] Sanchez E, Gutierrez-Carrasquilla L, Barbe F, Betriu A, Lopez-Cano C, Gaeta AM, Purroy F, Pamplona R, Ortega M, Fernandez E, Hernandez C, Lecube A, Simo R; ILERVAS Project. Lung function measurements in the prediabetes stage: data from the ILERVAS Project. Acta Diabetol. 2019 Sep;56(9):1005-1012. doi: 10.1007/s00592-019-01333-6. Epub 2019 Apr 15. PMID 30989377
- [Result] Sanchez E, Betriu A, Salas-Salvado J, Pamplona R, Barbe F, Purroy F, Farras C, Fernandez E, Lopez-Cano C, Mizab C, Lecube A; ILERVAS project investigators. Mediterranean diet, physical activity and subcutaneous advanced glycation end-products' accumulation: a cross-sectional analysis in the ILERVAS project. Eur J Nutr. 2020 Apr;59(3):1233-1242. doi: 10.1007/s00394-019-01983-w. Epub 2019 May 7. PMID 31065845
- [Result] Sanchez M, Sanchez E, Hernandez M, Gonzalez J, Purroy F, Rius F, Pamplona R, Farras-Salles C, Gutierrez-Carrasquilla L, Fernandez E, Bermudez-Lopez M, Salvador J, Salas-Salvado J, Lecube A; ILERVAS project collaborators. Dissimilar Impact of a Mediterranean Diet and Physical Activity on Anthropometric Indices: A Cross-Sectional Study from the ILERVAS Project. Nutrients. 2019 Jun 17;11(6):1359. doi: 10.3390/nu11061359. PMID 31212934
- [Derived] Leon-Mengibar J, Malagon MM, Bermudez-Lopez M, Valdivielso JM, Pamplona R, Torres G, Mauricio D, Castro E, Fernandez E, Caixas A, Hernandez M, Lopez-Cano C, Gordon A, Guzman-Ruiz R, Cusi K, Lecube A. Association of estimated liver fibrosis with carotid but not femoral atherosclerotic burden: the ILERVAS cohort. Front Endocrinol (Lausanne). 2026 Jan 6;16:1651689. doi: 10.3389/fendo.2025.1651689. eCollection 2025. PMID 41567808
- [Derived] Leon-Mengibar J, Bermudez-Lopez M, Valdivielso JM, Pamplona R, Torres G, Mauricio D, Castro-Boque E, Fernandez E, Caixas A, Bueno M, Ciudin A, Hernandez M, Simo R, Hernandez C, Lecube A. Impact of the new EASO obesity definition on the detection of atheromatosis in subjects with low-to-moderate cardiovascular risk. Front Endocrinol (Lausanne). 2025 Oct 10;16:1689960. doi: 10.3389/fendo.2025.1689960. eCollection 2025. PMID 41141356
- [Derived] Bermudez-Lopez M, Marti-Antonio M, Castro-Boque E, Bretones MDM, Farras C, Torres G, Pamplona R, Lecube A, Mauricio D, Valdivielso JM, Fernandez E. Development and Validation of a Personalized, Sex-Specific Prediction Algorithm of Severe Atheromatosis in Middle-Aged Asymptomatic Individuals: The ILERVAS Study. Front Cardiovasc Med. 2022 Jul 14;9:895917. doi: 10.3389/fcvm.2022.895917. eCollection 2022. PMID 35928938
- [Derived] Bermudez-Lopez M, Martinez-Alonso M, Castro-Boque E, Betriu A, Cambray S, Farras C, Barbe F, Pamplona R, Lecube A, Mauricio D, Purroy F, Valdivielso JM, Fernandez E; ILERVAS project collaborators. Subclinical atheromatosis localization and burden in a low-to-moderate cardiovascular risk population: the ILERVAS study. Rev Esp Cardiol (Engl Ed). 2021 Dec;74(12):1042-1053. doi: 10.1016/j.rec.2020.09.015. Epub 2020 Nov 6. English, Spanish. PMID 33162389
- [Derived] Sanchez E, Betriu A, Lopez-Cano C, Hernandez M, Fernandez E, Purroy F, Bermudez-Lopez M, Farras-Salles C, Barril S, Pamplona R, Rius F, Hernandez C, Simo R, Lecube A; ILERVAS project collaborators. Characteristics of atheromatosis in the prediabetes stage: a cross-sectional investigation of the ILERVAS project. Cardiovasc Diabetol. 2019 Nov 15;18(1):154. doi: 10.1186/s12933-019-0962-6. PMID 31729979
- See also: Study website — http://www.elbusdelasalut.cat/